CLINICAL TRIAL: NCT03999255
Title: REDUCING KIDNEY MOTION: OPTIMIZING ANESTHESIA AND COMBINING RESPIRATORY SUPPORT FOR RETROGRADE INTRARENAL SURGERY: A PILOT STUDY
Brief Title: SEARCH FOR OPTIMAL ANAESTHESIA IN RETROGRADE INTRARENAL SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, nariman.gadjiev, Head of Endourology, St. Petersburg State Pavlov Medical University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: №3/18
Record Dates: First submitted 2019-06-23; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing intrarenal surgery (Experimental)
  Interventions: Procedure: combined respiratory support (CRS)

INTERVENTIONS:
Procedure: combined respiratory support (CRS) — combined respiratory support (CRS) which consisted of reduction of tidal volume to 250-300 ml and respiratory rate to 4-5 per minute with transcatheter high-frequency jet ventilation (HFJV) through an endotracheal tube with a respiratory cycle frequency (RCF) of 300 per minute and maintained during RIRS.

SUMMARY:
Patients undergoing retrograde intrarenal surgery for kidney stones from November 2017 to May 2018 were prospectively recruited to participate in the study. In each case after the beginning of general anesthesia with mechanical ventilation surgeons were asked to assess the mobility of the operative field and conditions for laser lithotripsy according to the developed questionnaire scale. The questionnaire consisted of 5 degrees of assessment of kidney mobility and each question was scored from 1 to 5, 1 being very mobile (extremely poor conditions for dusting) and 5 completely immobile (Ideal conditions for dusting). After this assessment modified technique of general anesthesia was applied called combined respiratory support which consisted of reduction of tidal volume to 250-300 ml and respiratory rate to 4-5 per minute with transcatheter high frequency jet ventilation through endotracheal tube with a respiratory cycle frequency of 300 per minute and maintained during retrograde intrarenal surgery. At the beginning of combined respiratory approach, surgeons were once again asked to assess the mobility of the operative field and the conditions for laser lithotripsy. Main ventilation parameters were recorded and compared in both regimens.

ELIGIBILITY:
Inclusion Criteria:

* Kidneys stones with indications for retrograde intrarenal surgery

Exclusion Criteria:

* Patients with ASA class of greater than 3
* Patients with active urinary tract infection were excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Kidney motion assessed by the endourologist during retrograde intrarenal surgery | duration of RIRS Surgery
  a questionnaire was implemented in order to assess surgeon's feedback on novel technique. This was done in 2-step fashion in every patient and each patient served his own control: first, after the beginning of GA with MV in the mode of normal ventilation the questionnaire was implemented and surgeons were asked to assess the mobility of the operative field and the decency of conditions for laser lithotripsy.
  Second, novel CRS technique was then instituted and maintained throughout RIRS. Before lithotripsy itself surgeons were once again asked to assess the mobility of the operative field and conditions for laser lithotripsy according to the previously mentioned questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov Saint Petersburg Universuty, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gadzhiev N, Oibolatov U, Kolotilov L, Parvanyan S, Akopyan G, Petrov S, Cottone CM, Sung J, Okhunov Z. Reducing kidney motion: optimizing anesthesia and combining respiratory support for retrograde intrarenal surgery: a pilot study. BMC Urol. 2019 Jul 5;19(1):61. doi: 10.1186/s12894-019-0491-3. PMID 31277626